CLINICAL TRIAL: NCT07276152
Title: Plasma Oxytocin Changes in Response to Music Modified by Sonic Augmentation Technology vs Unaugmented Control Music in Healthy Controls and Patients With AVP-Deficiency
Brief Title: Plasma Oxytocin Changes in Response to Music Modified by Sonic Augmentation Technology
Acronym: TechnOXY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-01817, kt25christcrain6
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Sonic Augmentation Technology
Keywords: Arginine Vasopressin Deficiency; oxytocin; diabetes insipidus
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: Part 1 is a double-blinded, randomized and cross-over proof-ofconcept trial Part 2 is an open-labeled single arm pilot study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sonic augmentation technology (SAT) - placebo music (Experimental): Participants will listen to music enhanced with SAT in their first study visit. After a washout-phase of at least 20 hours they will come to a second study visit and they will listen to placebo music
  Interventions: Other: sonic augmentation technology
- placebo music- sonic augmentation technology (SAT) music (Experimental): Participants will listen to placebo in their first study visit. After a washout-phase of at least 20 hours they will come to a second study visit and they will listen to music enhanced with SAT
  Interventions: Other: sonic augmentation technology
- Sonic augmentation technology (SAT) in patients (Experimental): Patients have one study visit listening to SAT
  Interventions: Other: sonic augmentation technology

INTERVENTIONS:
Other: sonic augmentation technology — Participants/ patients listen to music enhanced with sonic aumentation technology

SUMMARY:
The investigator aim to investigate wheather music modified by sonic augmentation technology can produce increasing oxytocin levels with minimal to no side effects in a highly standardized setting

ELIGIBILITY:
Part 1:

Inclusion Criteria:

* Adult healthy controls
* No medication, except hormonal contraception

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Illicit substance use (except for cannabis) more than 10 times in lifetime or any time within the previous two months
* Consumption of alcoholic beverages >15 drinks/week
* Tobacco smoking >10 cigarettes/day
* Current or previous major psychiatric disorder (e.g., major depression, schizophrenia spectrum disorder)
* Psychotic disorder in first-degree relatives
* Pregnancy and breastfeeding

Part 2:

Inclusion Criteria:

* Confirmed diagnosis of AVP-Deficiency
* Age ≥ 18 years

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Illicit substance use (except for cannabis) more than 10 times in lifetime or any time within the previous two months
* Consumption of alcoholic beverages >15 drinks/week
* Tobacco smoking >10 cigarettes/day
* Current or previous major psychiatric disorder (e.g., major depression, schizophrenia spectrum disorder)
* Psychotic disorder in first-degree relatives
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in oxytocin levels in healthy adults after listening to SAT enhanced music vs. placebo music | up to 30 min
  Oxytocin release in response to music enhanced with SAT in healthy participants compared to oxytocin release in response to placebo stimulation in healthy participants
Change in oxytocin levels in patients with AVP-deficiency after listening to SAT enhanced music | up to 30 minutes
  baseline is defined as 100% of the initial value, in patients with AVP-Deficiency. Any changes will be expressed as a percentage relative to this baseline. Maximum oxytocin level observed between baseline and 30 minutes will be determined.

SECONDARY OUTCOMES:
Area under the concentration time curve in plasma oxytocin | up to 30 minutes
  will be assessed for music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Peak change in plasma oxytocin | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Time course of plasma oxytocin levels | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Time course of plasma copeptin | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Time course of plasma cortisol | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Time course of plasma neurophysin-1 | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Time course of other pituitary hormones/biomarkers | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT
Subjective/emotional effects assessed on numeric rating scale (NRS) | up to 30 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 30 min after listening to SAT.
  NRS will be presented as a range from 0 to 10 marked with "not at all" on the left and "extremely" on the right. The following NAS will be used: "any effect", "good effect", "bad effect", "liking", "high", "happy", "fear", "stimulated", "feeling close to others", "concentration", "thinking", "open", "trust", "want to be with other people", "loss of sense of time", and "the boundaries between myself and my surroundings seemed to blur".
Anxiety level using State-Trait Anxiety Inventory (STAI - State) | up to 35 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency. Baseline (before lisening to SAT) to 35 min after listening to SAT.
  Based on responses to 20 items, with scores ranging from 1 ("almost never") to 4 ("almost always"), a total score is calculated. The total trait score (STAI-T) ranges from 20 to 80, with higher scores indicating more pronounced anxiety and scores.
Frequency of specific body stress reactions using the Body Perception Questionnaire Short Form (BPQ-SF) | up to 50 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 50 min after listening to SAT.
  The BPQ-SF will be used to assess the frequency of specific body stress reactions in organs that are innervated by the autonomic nervous system (ANS).
  This study uses the Short Form (SF), totaling 46 items ranked from 1 (Never) to 5 (Always) to measure the frequency of specific body stress reactions. Though each unique part of the body may have its own reason for activation, the parts are linked by the ANS, a brain-body network that responds to everyday stress. Combined scores from organs throughout the body provide a measure of autonomic stress response patterns.
Recognition of emotions and body expressions in the EmBody/EmFace task | up to 35 minutes
  will be assessed music enhanced with SAT compared to placebo music in healthy adults and for music enhanced with SAT in patients with AVP-Deficiency Baseline (before lisening to SAT) to 35 min after listening to SAT.
  The EmBody and EmFace subtasks comprise each of 42 stimuli showing body or facial expressions of angry, happy, or neutral affect (14 clips per emotion, half in front view and half in half-profile side view from the left). Stimuli last 1.5 seconds at 24 frames per second and are geometrically and optically standardized to prevent biases induced by ethnic cues (e.g., hair or skin tone) or clothing. Item order is pseudorandom to prevent sequence effects and was determined using the following constraints: the same emotion is shown no more than twice in a row; the same view per emotion is not shown consecutively (i.e., no angry-front, angry-front).
Assessment of blood pressure | up to 40 minutes
  safety assessment of systolic and diastolic blood pressure. Safety outcomes will be summarized using descriptive statistics.
Assessment of heart rate | up to 40 minutes
  Saftey assessment of heart rate. Safety outcomes will be summarized using descriptive statistics.
Assessment of body temperature | up to 40 minutes
  Safety assessment of body temperature. Safety outcomes will be summarized using descriptive statistics.
Assessment of plasma potassium | up to 30 minutes
  Safety assessment of plasma potassium. Safety outcomes will be summarized using descriptive statistics
Assessment of plasma sodium | up to 30 minutes
  Safety assessment of plasma sodium. Safety outcomes will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland